CLINICAL TRIAL: NCT06254703
Title: Venous Excess and Lung Ultrasound During Continuous Kidney Replacement Therapy in Critically Ill Patients (VExLUS-KRT)
Brief Title: Venous Excess and Lung Ultrasound During Continuous Kidney Replacement Therapy in Critically Ill Patients
Acronym: VExLUS-KRT
Status: Active, not recruiting | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nuttha Lumlertgul, MD, Principal investigator, Chulalongkorn University
Other Study IDs: 0899/66
Record Dates: First submitted 2024-01-28; First posted 2024-02-12 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Failure Stage 3
Keywords: Acute kidney injury; VexLUS; Critically ill; Kidney replacement therapy; Continuous kidney replacement therapy; POCUS
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients receiving CKRT: 1. Adults (≥ 18 years of age)
  2. Admitted to ICU
  3. Plan to initiate CKRT by clinician's judgement
  Interventions: Diagnostic Test: VexLUS (venous excess lung ultrasound)

INTERVENTIONS:
Diagnostic Test: VexLUS (venous excess lung ultrasound) — IVC, hepatic veins (HVs), portal veins (PVs) and intrarenal veins (IRVs), and lung ultrasound
  Other Names: Bioelectrical impedence (BIA); N-terminal pro B-type natriuretic peptide (NT-proBNP)

SUMMARY:
Hemodynamic management of critically ill patients has long been focused on the arterial side of the vasculature by assessing adequate perfusion pressure. However, the venous pressure is also of critical importance. Venous congestion can occur in patients with right ventricular failure, pulmonary hypertension or fluid overload. Fluid overload has harmful effects to end organs causing acute kidney injury (AKI), lung edema, multiorgan dysfunction and death. Vice versa, AKI can aggravate fluid retention and inflammation. The measurement of venous pressure usually relies on central venous pressure (CVP) and inferior vena cava diameter (IVC). However, CVP measurement has been associated with measurement errors and has low accuracy in predicting fluid responsiveness. Moreover, IVC collapsibility or distensibility is a static parameter and is associated with subjective variability.

Multiorgan Point-of-Care ultrasound (POCUS) can enhance the management of AKI by enabling the evaluation of renal structural abnormalities and hemodynamic status . POCUS allows the clinician to assess intravascular and pulmonary fluid overload. It has been shown that POCUS is a good parameter to predict global fluid status of the patient .

Venous Excess Ultrasound (VEXUS) consists of the evaluation of IVC, hepatic vein, portal vein and intrarenal vein flow pattern. Previous studies showed significant correlation between VExUS score with RRT-free days and guide fluid management in critically ill patients with AKI . VExUS is useful in predicting patients at risk to develop AKI post cardiac surgery . Adding modified lung ultrasound score to the VExUS protocol could help clinician to adjust fluid administration and achieve proper fluid balance during continuous kidney replacement therapy (CKRT). However, the role of using combined VExUS and lung ultrasound in the assessment and guidance of fluid management during CKRT is unknown.

DETAILED DESCRIPTION:
Lung and cardiac ultrasonography can augment the definite diagnosis of volume overload. Thoracic ultrasound demonstrating B-lines which suggest thickened interstitial or fluid filled alveoli or increased vena cava diameter by ultrasound can also be used to assess volume status.

Recently, the venous excess ultrasound grading system (VExUS) has been introduced to be used in conjunction with POCUS to assess significant congestion. This technique used to classify the level of venous congestion by assessing the abdominal blood flow, including hepatic veins (HVs), portal veins (PVs) and intrarenal veins (IRVs). Abnormal patterns of flow in these organs can enhance the clinical evaluation of venous congestion in addition to Inferior vena cava (IVC) ultrasound since organ dysfunction occurring with venous congestion can also be from the transmission of pressure from right atrium (right atrial pressure, RAP) to the peripheral organ. Venous congestion is classified into four grades , ranging from grade 0 (no congestion) to the most severe form, grade 3 (severe congestion) or VExUS "A" through "E" Lung ultrasound and AKI Volume overload is associated with interstitial edema which increases the diffusion distance for oxygen and induces an increase in interstitial fluid pressure, impairing capillary blood flow and exacerbating organ dysfunction . A prospective pilot observational study with 45 adult patients with AKI at any time during ICU stay employed the FALLS (Fluid Administration Limited by Lung Ultrasound) protocol in which they use the LUS for assessing volume status. A new onset of the B-lines was considered as the endpoint of fluid administration. The study demonstrated a linear correlation between baseline B-line scores and PaO2/FiO2 ratio in ICU patients VExUS and lung ultrasound during CKRT

Previous studies have shown that VExUS and lung ultrasound may play a role in predicting AKI severity and may aid fluid de-escalation in critically ill patients. However, no studies have evaluated the role of both VExUS and lung ultrasound in guiding fluid management during CKRT. Our research aims to evaluate the prevalence of venous congestion by VExUS and lung ultrasound (VExLUS) during CKRT and its association with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years of age)
2. Admitted to ICU
3. Plan to initiate CKRT by clinician's judgement

Exclusion Criteria:

1. Refuse to participate
2. Previous diagnosis of end-stage kidney disease (ESKD) currently on kidney replacement therapy
3. Kidney tran splant recipient
4. Receive KRT before ICU admission
5. Structural kidney diseases which will interfere with intrarenal doppler ultrasound e.g. renal artery stenosis, autosomal dominant polycystic kidney disease etc.
6. Patients with previously known conditions that interfere with portal doppler assessment, namely liver cirrhosis, severe tricuspid regurgitation with structural heart disease or massive ascites.
7. Underlying disease process with a life expectancy less than 90 days
8. Pregnancy
9. Concomitant severe respiratory distress syndrome
10. Expected life expectancy <48 hours
11. Receiving extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients without ESRD that initiate CKRT
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of venous congestion by using VExLUS in patients who receive CKRT | 1 day
  prevalence of venous congestion

SECONDARY OUTCOMES:
To evaluate the association between VExLUS scores and all-cause mortality within 90 days, KRT-free days, ventilator-free days, vasopressor-free days, ICU-free days, dialysis dependence ay 28 days and 90 days | up to 90 days
  clinical outcomes
- to assess the correlation of VExLUS score with bioelectrical impedance vector analysis (BIVA) parameters and biomarkers | 1 day
  Correlation to BIVA
to evaluate inter-observer variability in determining VExLUS | 3 days
  inter-observer variability
To evaluate the association between VExLUS scores and all-cause mortality within 28 days | 28 days
  28 days all cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- King chula memorial hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No